CLINICAL TRIAL: NCT05722665
Title: The Predictive Capacity of a Convolutional Neural Network (CNN) Model to Detect Viral Pneumonia in Adult Patients With Coronavirus Disease 2019 (COVID-19) in Cali, Colombia
Brief Title: Convolutional Neural Network Model to Detect Coronavirus Disease 2019 (COVID-19) Pneumonia in Chest Radiographs
Acronym: RedNeumon
Status: Completed | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Universidad Autonoma de Occidente (Other)
Responsible Party: Sponsor
Other Study IDs: 1805
Record Dates: First submitted 2023-02-08; First posted 2023-02-10 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 (Coronavirus Disease 2019); COVID-19 Pneumonia
Keywords: COVID-19 (coronavirus disease 2019); Diagnostic Imaging; Radiography; Thorax; Computer Neural Network; Deep Learning
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal chest radiographs: X-rays without alterations in the lung parenchyma
  Interventions: Other: Categorization of chest xrays images
- COVID-19 chest radiographs: X-rays belonging to patients with a diagnosis of COVID-19 confirmed by positive Reverse Transcriptase polymerase chain reaction (RT-PCR) and/or presence of antibodies to COVID-19 and/or positive COVID-19 viral antigen.
  Interventions: Other: Categorization of chest xrays images
- Other pneumonia chest radiographs: X-rays belonging to patients with a diagnosis of pneumonia other than COVID-19
  Interventions: Other: Categorization of chest xrays images

INTERVENTIONS:
Other: Categorization of chest xrays images — Use of Convolutional Neural Network Model to categorize chest xrays images in each group.

SUMMARY:
This study aims to design a Convolutional Neural Network (CNN) and apply an attention model to help differentiate pneumonia due to Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), pneumonia due to other viruses/bacteria, and normal chest x-ray (CXR) in clinical practice. A bank of digital chest images from a high-complexity health facility in Cali, Colombia, was used.

DETAILED DESCRIPTION:
To differentiate coronavirus disease 2019 (COVID-19) pneumonia from other types of pneumonia, expert radiologists must analyze the chest x-ray (CXR) to identify visual, radiographic patterns associated with Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. It is challenging because the findings are similar for different types of pneumonia.

Since the manual diagnosis of COVID-19 from CXR is a difficult and time-consuming process, applying deep learning (DL) models to medical image analysis is a current hot research topic. This work will develop a new Convolutional Neural Network (CNN) to detect COVID-19 radiographs. It will use a large dataset of chest radiographs classified into three classes: viral/bacterial pneumonia, COVID-19 pneumonia, and normal images. The study aims to incorporate a new attention module that applies CNNs to the linear projection operation to help differentiate COVID-19 pneumonia from other pneumonia and normal chest radiographs in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiographs from patients without COVID-19 or other pneumonia took before the pandemic start date (January 2020)
* Chest radiographs from patients with COVID-19 confirmed by positive Reverse Transcriptase polymerase chain reaction (RT-PCR) and/or presence of antibodies to COVID-19 and/or positive COVID-19 viral antigen.
* Chest radiographs from patients without COVID-19 confirmed by a negative Reverse Transcriptase polymerase chain reaction (RT-PCR) and other pneumonia diagnoses taken before the pandemic start date (January 2020)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: X-rays without alterations in the lung parenchyma Group 2: X-rays belonging to patients with a diagnosis of pneumonia other than COVID-19 Group 3: X-rays belonging to patients with a diagnosis of COVID-19 confirmed by positive Reverse Transcriptase polymerase chain reaction (RT-PCR) and/or presence of antibodies to COVID-19 and/or positive COVID-19 viral antigen.
Sampling Method: Non-Probability Sample
Enrollment: 3599 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 (coronavirus disease 2019) pneumonia chest radiograph identified | month 8
  Development and determination of the predictive capacity of a Convolutional Neural Network model to detect viral pneumonia in chest radiographs of adult patients with acute respiratory disease secondary to SARS-COV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Fernandez, M.D, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No